CLINICAL TRIAL: NCT04381403
Title: Development of Toothpaste for the Removal of Dental Calculus: a Double-blind, Randomized Controlled Trial.
Brief Title: Development of a New Toothpaste for the Removal of Dental Calculus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faleh Tamimi (Other)
Collaborators: MedTeq (Industry); Mitacs (Industry); Visionaturolab INC. (Unknown); Cégep Garneau (Unknown)
Responsible Party: Sponsor-Investigator, Faleh Tamimi, Associate professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A08-M35-16B
Record Dates: First submitted 2020-04-30; First posted 2020-05-08 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Calculus, Dental; Periodontal Diseases; Periodontal Inflammation
Keywords: Oral Hygiene; Calculus; Dental plaque
MeSH Terms: conditions — Dental Calculus; Periodontal Diseases; Calculi; Dental Plaque

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bio-descaling D-Tart toothpaste (Experimental): Bio-descaling D -Tart is a bio-descaler toothpaste that is manufactured at Du-Var laboratories (1460 Graham Bell, Boucherville, Québec, Canada J4B 6H5)
  Interventions: Other: Bio-descaling D-Tart toothpaste
- Crest® (Active Comparator): anti-tartar toothpaste, Complete Whitening plus Scope, tartar control produced by Procter & Gamble, Cincinnati, OH),
  Interventions: Other: Crest® toothpaste

INTERVENTIONS:
Other: Bio-descaling D-Tart toothpaste — Patients received Bio-descaling D-Tart toothpaste, which is a new dentifrice (Visionaturolab Inc., QC) that contains a natural bio-descaler powder of cuttlefish bone
  Arms: Bio-descaling D-Tart toothpaste
Other: Crest® toothpaste — Patients received Crest toothpaste; Anti-tartar toothpaste
  Arms: Crest®

SUMMARY:
Periodontal disease is amongst the most prevalent oral diseases worldwide and in North America. According to the 2007/09 Canadian Health Measures Survey, 16% of Canadian adults and 24% of older adults, 60 to 79 years of age, were found to have moderate periodontal disease. Moreover, 11% of Canadian adults were found to have calculus scores in the highest range. On the other hand, recent reports on the prevalence of periodontitis in the US showed that 47.2% of adults aged 30 years and older have some form of periodontal disease and 70.1% of adults 65 years and older have periodontal disease. The estimates also showed that the expenditure for periodontal treatments in the US is about approximately $ 14.3 billion.

Since dental calculus plays an important etiological role in initiation and progression of periodontal diseases. Investigation and investment on preventive technologies to prevent the periodontal disease are important for any health care system and its end-users. Furthermore, the removal and prevention of dental calculus using an effective toothpaste could reduce the need for professional periodontal interventions or the time of these treatments that in turn reduces their cost and other burdens on patients.

The aim of this study is to assess the efficacy of D-Tart toothpaste in removing dental calculus compared to Crest® (Complete Whitening plus Scope, tartar control, Procter & Gamble, Cincinnati, OH), anti-tartar toothpaste with similar pH and texture to D- Tart toothpaste.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over, to ensure compliance with the study instructions
* Systemically healthy to exclude the possibility of calculus formation due to disease;
* Has at least 20 sound natural teeth including all lower anterior teeth, the main location of calculus build up;
* Having the history of previous calculus formation (at least 1.5 mm of calculus width) on the lingual surfaces of the mandibular anterior teeth after 3- 6 months of receiving a professional prophylaxis treatment, for better assessment of the toothpaste effectiveness;
* Agree to follow the study instruction: adherence to study arm, for the study timeline.

Exclusion Criteria:

* Pregnancy: pregnant women at high risk of developing gum inflammation that usually occurs during pregnancy, which could introduce bias to the study;
* any physical handicap, psychological or health conditions that might jeopardize the ability of the patient to brush his/ her teeth, these complications cause bias in the study;
* Antibiotics or anti-inflammatory drugs are taken within 1 month prior to the study, to avoid bias when assessing the gum health;
* Currently using Chlorhexidine oral products, since these products can affect biofilm and calculus formation, therefore they can introduce bias in our assessment of calculus removal by our toothpaste;
* Sensitivity to tartar-control toothpaste;
* Patients currently receiving dental treatment that would result in the removal of plaque or calculus and compromise our ability to measure calculus removed by the toothpaste;
* unable to return for evaluations/study recalls, to avoid the significant loss in the number of participants; 9) Having the diagnosis of Periodontal Screening and Recording scale (PSR) of 4, these type of patients have advanced periodontitis with a high risk of tooth loss (periodontal pockets of 6 mm and more) and could bias the treatment outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Change in calculus index | Baseline, 3 months, 9 months
  Calculus level in mm on teeth before and after brushing with toothpaste.

SECONDARY OUTCOMES:
Modified Gingival Index | Baseline, 3 months, 9 months
  semi-quantitative assessment of gingival health around each tooth
  Absence of inflammation; Mild inflammation or with slight changes in color and texture but not in all portions of gingival marginal or papillary
  Mild inflammation, such as the preceding criteria, in all portions of gingival marginal or papillary
  Moderate, bright surface inflammation, erythema, edema and/or hypertrophy of gingival marginal or papillary
  Severe inflammation: erythema, edema and/or marginal gingival hypertrophy of the unit or spontaneous bleeding, papillary, congestion or ulceration
Shaw and Murray Stain Index | baseline, 3 months, 9 months
  Quantitative assessment of extrinsic stains on the labial and palatal/lingual surfaces of the upper and lower central and lateral incisors; The outline of the labial and lingual surfaces of all eight incisor teeth are enlarged to scale (magnification X 4) and each tooth face divided into 4-mm squares. All areas of extrinsic stain are drawn by the examiner on a grid system and then measured.
Quigley-Hain plaque index (QHI) | baseline, 3 months, 9 months
  semi-quantitative assessment of plaque around each tooth;
  Score 0: No plaque Score 1: Isolated flecks of plaque at the gingival margin Score 2: A continuous band of plaque up to 1mm at the gingival margin Score 3: Plaque greater than 1mm in width and covering up to one third of the tooth surface Score 4: Plaque covering from one thirds to two thirds of the tooth surface Score 5: Plaque covering more than two thirds of the tooth surface

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Faculty of Dentistry, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
The research team will collect the personal information of participants. This may include their name, address, phone number, health plan number, date of birth, dental and medical history, and medical-related information, which shall be collected from all participants by asking them to fill dental and medical history forms. All information collected from participants will be kept Confidential at the study site and secure in a locked file cabinet in Cégep Garneau. The electronically stored information would be also secured in a computer hard drive accessible only to researchers with a confidential access code. This information will be kept for 5 years after the study is terminated. All study data will also be sent to the sponsor and/or its representatives, as long as they agree to use the information as described previously. However, this data will not identify the participants by name.